CLINICAL TRIAL: NCT06788197
Title: A Phase Ib/II Study of SHR-A1811 and Fulvestrant in Combination With or Without HS-10352 in Locally Advanced or Metastatic Breast Cancer Patients Who Progressed After Adjuvant Therapy
Brief Title: A Study of SHR-A1811 and Fulvestrant, With or Without HS-10352, in Locally Advanced or Metastatic Breast Cancer Patients
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Chief Physician, Henan Cancer Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-528
Record Dates: First submitted 2025-01-21; First posted 2025-01-23 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Locally Advanced or Metastatic Breast Cancer
Keywords: Breast Cancer; SHR-A1811; HS-10352
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: SHR-A1811 + fulvestrant group: SHR-A1811+fulvestrant ；
  HS-10352 group: SHR-A1811+Fulvestrant+HS-10352
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A1811 + fulvestrant group (Experimental): Subjects will receive SHR-A1811 combined with fulvestrant therapy.
  Interventions: Drug: SHR-A1811+ Fulvestrant
- HS-10352 group (Experimental): Subjects will receive SHR-A1811 combined with Fulvestrant and HS-10352 therapy.
  Interventions: Drug: SHR-A1811+ Fulvestrant+HS-10352

INTERVENTIONS:
Drug: SHR-A1811+ Fulvestrant — SHR-A1811 is administered intravenously; fulvestrant is administered Intramuscular
  Arms: SHR-A1811 + fulvestrant group
Drug: SHR-A1811+ Fulvestrant+HS-10352 — SHR-A1811 is administered intravenously; fulvestrant is administered Intramuscular ； HS-10351 is administered orally
  Arms: HS-10352 group

SUMMARY:
This study is being conducted to evaluate the efficacy and safety of SHR-A1811 and Fulvestrant in Combination with or without HS-10352 in locally advanced or metastatic breast cancer patients. Subjects will receive SHR-A1811 and Fulvestrant in Combination with or without HS-10352.

DETAILED DESCRIPTION:
This study plans to enroll breast cancer patients whose disease progressed during treatment or within 12 months of completing adjuvant therapy and who have not received prior systemic therapy. SHR-A1811 + fulvestrant group will receive treatment with SHR-A1811 and fulvestrant. HS-10352 group will receive treatment with SHR-A1811, fulvestrant, and HS-10352. Treatment will continue until disease progression or the occurrence of intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥18 years and ≤75 years;
2. ECOG Performance Status of 0 -2;
3. Locally advanced/metastatic breast cancer not amenable to curative therapy
4. Disease progression during treatment or within 12 months of completing adjuvant therapy ;
5. No prior anti-cancer systemic therapy has been administered;
6. Fasting blood glucose < 126 mg/dL, and HbA1C < 6.0%;
7. Life expectancy of ≥3 months;
8. Patients have at least one target lesion according to RECEST 1.1;
9. Adequate function of major organs;
10. Female patients who are either premenopausal or have not undergone surgical sterilization: during the treatment period and for at least 7 months after the final dose of study medication, agree to abstain from sexual activity or utilize effective contraceptive methods.
11. Sign Informed Consent Form.

Exclusion Criteria:

1. Breast cancer that has not been histologically confirmed;
2. Inflammatory breast cancer;
3. Participants ineligible for endocrine therapy due to any disease burden, as judged by the investigator;
4. Meningeal metastasis or active parenchymal brain metastasis;
5. Presence of diabetes symptoms, history of primary diabetes, gestational diabetes, steroid-induced diabetes, or other secondary diabetes;
6. Prior anti-cancer systemic therapy has been administered;
7. Use of investigational drugs within 4 weeks；
8. Received immunotherapy, macromolecular targeted therapy, or other antitumor biologics within 4 weeks; or received endocrine therapy, chemotherapy, small molecule targeted drug therapy, or traditional Chinese medicine treatment with antitumor indications within 2 weeks;
9. Received radical radiotherapy within 4 weeks, or received palliative radiotherapy within 2 weeks;
10. Previously received antitumor treatment or radiotherapy for any malignancy, excluding malignancies such as cured cervical carcinoma in situ, basal cell carcinoma, or squamous cell carcinoma;
11. A history of other malignancies within the past 5 years, excluding cured cases of skin basal cell carcinoma and cervical carcinoma in situ;
12. Prior anti-tumor treatment toxicities have not yet recovered to NCI CTCAE V5.0 grade ≤1 or baseline levels;
13. A history of immunodeficiency, including HIV positivity, other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
14. Interstitial pneumonia/interstitial lung disease, or presence of moderate to severe pulmonary disease that may interfere with the detection or management of drug-related pulmonary toxicity within 3 months prior to the first administration of the study drug, as well as any autoimmune, connective tissue, or inflammatory diseases involving the lungs, or a history of total pulmonary resection surgery
15. Presence of active hepatitis B, hepatitis C, liver cirrhosis, or severe infections requiring control with antibiotics, antiviral drugs, or antifungal medications;
16. History of hereditary or acquired bleeding and thrombotic tendencies (such as haemophilia, coagulation disorders, etc.);
17. Inability to swallow, intestinal obstruction, or the presence of other factors affecting drug intake and absorption;
18. Patients with known allergies or contraindications to the study drug and its excipient components;
19. Female patients who are pregnant or lactating, those of reproductive potential with a positive baseline pregnancy test, or those of reproductive age who are unwilling to use effective contraceptive measures throughout the entire study period;
20. According to the investigator's judgment, patients with severe concomitant diseases that pose a risk to their safety or prevent them from completing the study, a history of definite neurological or psychiatric disorders, including epilepsy or dementia, or any other condition deemed by the investigator to make the patient unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 52 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) according to RECIST1.1 （SHR-A1811+fulvestrant group and HS-10352 group (Phase II)） | Up to approximately 4 years
  ORR defined as the proportion of patients with the best overall response of complete response or partial response，as determined by the investigator according to RECIST v1.1
Recommended Phase 2 dose (RP2D) (HS-10352 group (Phase Ib)) | From the first dose to the last dose of the first cycle defined as 28 days

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) （SHR-A1811 + fulvestrant group and HS-10352 group (Phase II)） | Up to approximately 4 years
  Evaluate the incidence and severity of adverse events according to CTCAE 5.0
Objective Response Rate (ORR) according to RECIST1.1 （HS-10352 group(Phase Ib)） | Up to approximately 4 years
  ORR defined as the proportion of patients with the best overall response of complete response or partial response，as determined by the investigator according to RECIST v1.1
Progression-Free Survival (PFS)（SHR-A1811 +fulvestrant group and HS-10352 group (Phase Ib/Phase II)） | Up to 4 years
  PFS is defined as the time from the first therapeutic dose to death or disease progression
Overall Survival (OS) （SHR-A1811 +fulvestrant group and HS-10352 group (Phase Ib/Phase II)） | Up to 4 years
  OS is defined as the time from the first therapeutic dose to death from any cause
Clinical Benefit Rate (CBR) （CR+ PR+ SD≥24weeks）（SHR-A1811 +fulvestrant group and HS-10352 group (Phase Ib/Phase II)） | Up to 4 years
  CBR is defined as the percentage of participants with a CR, PR, and/or stable disease (SD) for at least 24 weeks, as determined by the investigator according to RECIST v1.1
Duration of Response (DOR) （SHR-A1811 +fulvestrant group and HS-10352 group (Phase Ib/Phase II)） | Up to 4 years
  DOR is defined as the time from the first occurrence of a CR or PR to the first occurrence of disease progression as determined by the investigator according to RECIST v1.1, or death from any cause (whichever occurs first)

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhen Liu, MD, Principal Investigator — Henan Cancer Hospital

IPD SHARING:
Plan to Share IPD: No